CLINICAL TRIAL: NCT02101138
Title: An Open-Label, Proof-of-Concept Study to Evaluate the Safety and Efficacy of Dexpramipexole (KNS-760704) in Subjects With Hypereosinophilic Syndrome
Brief Title: Study to Evaluate Safety and Efficacy of Dexpramipexole (KNS-760704) in Subjects With Hypereosinophilic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140063; 14-I-0063
Record Dates: First submitted 2014-03-14; First posted 2014-04-02 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12-01

CONDITIONS: Hypereosinophilic Syndrome
Keywords: Corticosteroids; Eosinophilia
MeSH Terms: conditions — Hypereosinophilic Syndrome; Eosinophilia | interventions — Dexpramipexole

ARMS (1):
- Dexpramipexole (Experimental): Dexpramipexole treatment
  Interventions: Drug: Dexpramipexole

INTERVENTIONS:
Drug: Dexpramipexole — Dexpramipexole (KNS 760704) is a synthetic amino-benzothiazole developed for use in amyotrophic lateral sclerosis (ALS)

SUMMARY:
Background:

- Eosinophils are white blood cells that fight infections. In people with hypereosinophilic syndrome (HES), eosinophil levels are too high and can damage their organs. HES is usually treated with steroids, but steroids can cause side effects and stop working over time. Researchers want to see if a drug called dexpramipexole, being developed by Knopp Pharmaceuticals, can help people with HES to reduce their steroid dose.

Objective:

- To test whether dexpramipexole can reduce the steroid dose needed to control eosinophilia and HES symptoms.

Eligibility:

- Adults 18 and older with HES who respond to steroids, but need more than 10 mg daily to control eosinophilia and symptoms.

Design:

* The study will last 9 months with 6 visits to NIH.
* Participants will be screened with medical history, physical exam, and urine and blood samples.
* Participants steroids will be tapered to the lowest effective dose. During this time, blood will be drawn weekly. Participants will take this dose for 2 weeks before starting the study drug.
* Participants will take the study drug twice daily by mouth for 12 weeks along with steroids. The steroid dose will not be decreased during this time and participants will be seen monthly for a medical history, physical examination and blood work.
* Just before and 12 weeks after starting the study drug, the following tests will be performed:
* medical history and physical exam
* blood and urine tests
* lung function tests
* electrocardiogram (measures heart electrical activity)
* echocardiogram (takes pictures of the heart using sound waves)
* bone marrow biopsy (a needle inserted into the hip bone that removes bone marrow cells for study)
* After 12 weeks, the participants steroid dose will be tapered again to the lowest effective dose while on study drug.
* Two weeks after the lowest effective dose is reached, participants will return for a medical history, physical examination, blood work, lung and heart tests.
* Participants who respond to the study drug may be able to continue to receive the drug on a planned separate study.
* Four weeks after stopping the study drug, participants will have medical history, physical exam, and blood tests.

DETAILED DESCRIPTION:
Hypereosinophilic syndromes (HES) are a heterogeneous group of disorders characterized by peripheral eosinophilia and evidence of eosinophil-related end organ damage. Although a high proportion of patients respond initially to corticosteroid therapy, high doses are often necessary to control the eosinophilia and clinical symptoms, and many patients become relatively refractory to therapy and/or develop serious side effects.

Dexpramipexole (KNS 760704) is a synthetic aminobenzothiazole shown to safely reduce blood eosinophils counts in individuals with amyotrophic lateral sclerosis (ALS) in several clinical trials. The purpose of this proof-of- concept study is to evaluate the effect of dexpramipexole, an orally bioavailable small molecule, on circulating and tissue eosinophils in 10 subjects with HES. Following completion of eligibility assessments, subjects with absolute eosinophil count (AEC) < 1000/uL will enter a lead-in period, during which a standardized weekly corticosteroid taper will be undertaken to establish a "minimally effective corticosteroid dose" in each study subject. For subjects whose symptoms are stable but AEC > 1000/uL at the time of enrollment, the steroid dose at the time of enrollment will be defined as the minimally effective corticosteroid dose and no taper will be performed. Once the minimally effective corticosteroid dose is established, treatment with dexpramipexole 150 mg twice daily will begin. A standardized corticosteroid taper will begin after 12 weeks of treatment with dexpramipexole to determine the "minimally effective corticosteroid dose on dexpramipexole". Eosinophil counts and routine chemistries will be monitored weekly during corticosteroid tapering. End organ assessment, including echocardiogram, pulmonary function testing, and other studies as appropriate will be performed at study baseline, initiation of dexpramipexole therapy, 3 months after initial dosing with dexpramipexole, and the end of study visit. Bone marrow assessment will be performed prior to and after 12 weeks of dexpramipexole. Drug levels will be assessed prior to dexpramipexole and at week 12 and week 24 of dosing.

The primary efficacy endpoint will be the number of subjects with a greater than or equal to 50 % change in prednisone (or equivalent) dose to maintain absolute eosinophil count (AEC) at or below baseline (pre-enrollment) levels and control clinical symptoms (responder analysis). Assuming that 10 patients received study drug per protocol, at least 4 of them will need to meet this endpoint to significantly show (at the usual two-sided 5% level, equivalent to the onesided 2.5% level) that at least 10% of patients respond to dexpramipexole (exact binomial test). Safety will be assessed as the incidence of adverse events (AEs) (including serious adverse events [SAEs]), vital signs, clinical laboratory assessments, physical examination, electrocardiogram (ECG) tests, and body weight. Exploratory endpoints will include determination of the effect of dexpramipexole on measures of eosinophil activation, cytokine/chemokine profile and other immunologic parameters, and reduction of tissue eosinophils.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject will be eligible for participation in the study only if all of the following criteria apply:

1. The subject is male or female, age greater than or equal to 18 years
2. The subject has a documented history of HES requiring greater than or equal to 10 mg prednisone (or equivalent) to maintain disease control.

   HES is defined as 1) peripheral blood eosinophilia (>1500 eosinophils/microL) on at least two occasions, 2) signs and symptoms of organ system involvement attributable to the eosinophilia, and 3) exclusion of secondary causes of eosinophilia, such as parasitic helminth infection, drug hypersensitivity and neoplasms, for which appropriate therapy is directed at the underlying cause
3. HES symptoms are stable on the current corticosteroid dose.
4. The subject agrees to storage of samples for study.
5. Females are eligible for this study if they are:

(1) of non-childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal as defined by no menses in 1 year); OR

(2) of childbearing potential but willing to practice effective contraception or abstinence during administration of the study drug and for 3 months after administration of the investigational study drug (dexpramipexole).

Participation of Women:

Contraception: Pre-clinical animal data demonstrated some fetal risk, suggesting there may a human reproductive risk. Subjects must agree not to become pregnant. Females of childbearing potential must have a pregnancy test before the first dose of dexpramipexole. Because of the risk involved, subjects and their partners must use two methods of birth control. They must continue to use both methods for 3 months after stopping the study drug. Two methods of birth control may be selected from the list included below:

* Hormonal contraception
* Male or female condoms with or without a spermicide
* Diaphragm or cervical cap with a spermicide
* Intrauterine device (IUD)

If pregnancy is suspected or should occur, subjects must notify the study staff immediately.

EXCLUSION CRITERIA:

A subject will not be eligible to participate in the study if any of the following conditions are fulfilled at the time of enrollment:

1. Life-threatening HES or other condition that, in the Investigator s opinion, places the subject at undue risk by participating in the study
2. Pregnant or breast-feeding
3. History of malignancy, including solid tumors and hematologic malignancies (except basal cell and squamous cell cancers of the skin that have been completely excised and cured)
4. HIV infection or any other known immunodeficiency.
5. Biopsy-proven eosinophilic granulomatosis with polyangiitis
6. Positive test for FIP1L1/PDGFRA fusion gene
7. Absolute neutrophil count <2000/microL at screening, or any documented history of neutropenia
8. Renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) of less than or equal to 80 mg/dL at screening (estimation of creatinine clearance using the MDRD formula).
9. Cardiac abnormality defined as:

   1. Moderate to severely decreased cardiac function (left ventricular ejection fraction (LVEF) < 20% or history of LVEF <20% within the past 6 months or NYHA class IIIb or IV)
   2. History of angina or acute myocardial infarction in the past 6 months
   3. History or long QT syndrome or arrhythmia.
   4. A prolongation of QT/QTc interval (e.g., repeated demonstration of a QT/QTc interval >450 ms before study treatment administration) at screening, admission or pre-dose on Day 1.
   5. Any clinically important abnormalities in resting ECG that may interfere with the interpretation of QTc interval changes at screening, admission or pre-dose on Day 1.

   This includes subjects with any of the following:

   i. PR interval >210 ms;

   ii. QRS >110 ms;

   iii. Heart rate <45 bpm or >100 bpm (average of 3 assessments).
10. Recent history or suspicion of drug or alcohol abuse in the preceding 6 months
11. Treatment with an investigational drug in the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03-14; Primary Completion 2016-12-30 (Actual); Study Completion 2019-10-23 (Estimated)

PRIMARY OUTCOMES:
The corticosteroid dose after treatment with 150 mg twice daily of dexpramipexole as a percentage of the corticosteroid dose prior to treatment | After 3 months of taking dexpramipexole
The number of subjects with a greater than or equal to 50 % change in prednisone (or equivalent) dose to maintain absolute eosinophil count (AEC) at or below baseline (pre-enrollment)levels and control clinical symptoms | After 3 months of taking dexpramipexole

SECONDARY OUTCOMES:
Reduction in circulating eosinophil and bone marrow eosinophil count after 3 months of treatment with dexpramipexole (prior to steroid taper) | After 3 months of dexpramipexole therapy
The number of subjects able to taper to <10 mg prednisone (or equivalent) dose to maintain absolute eosinophil count (AEC) at or below baseline (pre-enrollment) levels and control clinical symptoms | After 3 months of dexpramipexole therapy
Incidence and severity of adverse events | During dexpramipexole therapy

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Klion, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ogbogu PU, Bochner BS, Butterfield JH, Gleich GJ, Huss-Marp J, Kahn JE, Leiferman KM, Nutman TB, Pfab F, Ring J, Rothenberg ME, Roufosse F, Sajous MH, Sheikh J, Simon D, Simon HU, Stein ML, Wardlaw A, Weller PF, Klion AD. Hypereosinophilic syndrome: a multicenter, retrospective analysis of clinical characteristics and response to therapy. J Allergy Clin Immunol. 2009 Dec;124(6):1319-25.e3. doi: 10.1016/j.jaci.2009.09.022. PMID 19910029
- [Background] Bozik ME, Mather JL, Kramer WG, Gribkoff VK, Ingersoll EW. Safety, tolerability, and pharmacokinetics of KNS-760704 (dexpramipexole) in healthy adult subjects. J Clin Pharmacol. 2011 Aug;51(8):1177-85. doi: 10.1177/0091270010379412. Epub 2010 Oct 19. PMID 20959524
- [Background] Cudkowicz ME, van den Berg LH, Shefner JM, Mitsumoto H, Mora JS, Ludolph A, Hardiman O, Bozik ME, Ingersoll EW, Archibald D, Meyers AL, Dong Y, Farwell WR, Kerr DA; EMPOWER investigators. Dexpramipexole versus placebo for patients with amyotrophic lateral sclerosis (EMPOWER): a randomised, double-blind, phase 3 trial. Lancet Neurol. 2013 Nov;12(11):1059-67. doi: 10.1016/S1474-4422(13)70221-7. Epub 2013 Sep 23. PMID 24067398
- [Derived] Panch SR, Bozik ME, Brown T, Makiya M, Prussin C, Archibald DG, Hebrank GT, Sullivan M, Sun X, Wetzler L, Ware J, Fay MP, Dunbar CE, Dworetzky SI, Khoury P, Maric I, Klion AD. Dexpramipexole as an oral steroid-sparing agent in hypereosinophilic syndromes. Blood. 2018 Aug 2;132(5):501-509. doi: 10.1182/blood-2018-02-835330. Epub 2018 May 8. PMID 29739754
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-I-0063.html